CLINICAL TRIAL: NCT06085404
Title: Patients Derived Organoids (PDOs) Immune Cells Co-culture in Ovarian Cancer: the Role of TUmoR microEnvironment.
Brief Title: Patients Derived Organoids in Ovarian Cancer
Acronym: PICTURE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4531
Record Dates: First submitted 2023-06-21; First posted 2023-10-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Participants are prospectively assigned to an intervention consisting of a blood draw and tumor biopsy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Other): Participants are prospectively assigned to an intervention consisting of a blood draw and tumor biopsy.
  Interventions: Procedure: Blood sample

INTERVENTIONS:
Procedure: Blood sample — Patients will be enrolled starting right after Ethics Committee approval. Samples will be taken during surgery that will take place in the operating rooms of oncological gynecology.
  Other Names: Tumor Biopsy

SUMMARY:
Among cancer models, patients derived organoids (PDOs) best reproduce tumor's tissue architecture, intratumor heterogeneity and are able to mimic in vivo patients' drugs response.

For these reasons, it has been designed a study to assess the feasibility of PDOs immune cells co-culture in OC patients and the concordance between ex vivo sensitivity and in vivo treatment response. If proven effective and reliable, PDOs could be introduced into clinical practice as empirical predictor of patients' response to antineoplastic drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Preoperative clinical, serological and radiologic suspicion of International Federation of Gynecology and Obstetrics (FIGO) stage IIIC or greater ovarian, fallopian tube, or primary peritoneal cancer;
2. Histologic diagnoses of epithelial ovarian cancer at frozen section
3. Age >18 and years;
4. Estimated life expectancy of at least 4 weeks;
5. Performance status (PS) according to Eastern Cooperative Oncology Group (ECOG) < 2

Exclusion Criteria:

1. Non-serous histology at frozen section;
2. Patients with a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (> 10 mg equivalent prednisone/daily) or any other form of immunosuppressive therapy within 7 days prior to the enrollment.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-11-25 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
To improve the knowledge of advanced ovarian cancer by developing an experimental laboratory model. | 24 months
  To improve the knowledge of advanced ovarian cancer by developing an experimental laboratory model, organoids, aimed at obtaining information on the genomic and molecular characteristics of tumor cells and cells belonging to the immune system specific to each individual ovarian cancer patient and to study their interaction.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Nero, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Policlinico Universitario Agostino Gemelli, Roma, Italy

IPD SHARING:
Plan to Share IPD: No